CLINICAL TRIAL: NCT07001371
Title: Emotional Brain Training for Addiction Medicine Treatment - A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: University of California, San Francisco (Other); Social Action for Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000383
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Use Disorder; Stimulant Use Disorder; Opioid Use Disorder; Tobacco Use Disorder; Alcohol Use Disorder; Sedative, Hypnotic, or Anxiolytic Use Disorders
Keywords: early remission; sustained remission
MeSH Terms: conditions — Opioid-Related Disorders; Tobacco Use Disorder; Alcoholism

STUDY DESIGN:
Intervention Model Description: Randomized 8 weeks of Standard of Care (SOC) addiction treatment versus SOC plus Emotional Brain Training (EBT).
  Subjects are patients currently receiving SOC at the Addiction Recovery Clinic at SAC Health. As part of SOC, participants will complete the Brief Addiction Monitor (BAM) tool at weeks 0, 4, and 8, and the Adverse Childhood Events (ACES) survey at week 0.
  Providers at the clinic will approach subjects regarding participation in the study.
  Subjects randomized to the EBT arm will receive 8 weeks of the standard EBT intervention, which includes:
  Subjects randomized to the control arm, in addition to SOC, will have access to:
  * Individual case management services
  * Drug and alcohol counseling
  * The opportunity to transition to the EBT arm after completion of two months in the control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Participants will receive SOC, which includes medications for addiction therapy (MAT) (including but not limited to buprenorphine, naltrexone, bupropion, etc.) weekly counseling, and monthly clinic visits with addiction specialists.
  Interventions: Other: Standard addiction counseling and medical therapy
- Emotional Brain Training (EBT) and Standard of Care (SOC) (Experimental): This group will receive all the components of SOC plus EBT counseling:
  A. The components below will be completed daily and is estimated to take 25 minutes:
  i. [10 1-minute spiral ups (SU) - an EBT specific, app-directed methodology of emotional regulation], plus; ii. 5 minutes via telephone for a group peer connection iii. 10 minutes online/phone app coursework/video
  B. Once a week: participants will participate in a 60 minute small-group telephone meeting for accountability and support C. Once a week: participants will participate in at least 3 30-minute Spiral Up (SU) groups/week to practice the skills. These are available online daily.
  Interventions: Behavioral: Emotional Brain Training; Other: Standard addiction counseling and medical therapy

INTERVENTIONS:
Behavioral: Emotional Brain Training — Emotional Brain Training (EBT) is a structured, neuroscience-based behavioral intervention that focuses on rewiring the brain's stress-related circuits to promote emotional resilience, self-regulation, and lasting behavioral change. This behavioral intervention has not been implemented in addiction treatments in the past. Unlike traditional therapies that primarily target cognitive processes or symptom management, EBT directly addresses the physiological and emotional root causes of maladaptive behaviors by engaging the brain's natural neuroplasticity mechanisms. EBT integrates rapid emotional processing tools, peer-to-peer support, clinician-facilitated sessions, and mobile app-based self-care to systematically transition brain circuits from stress-reactive to stress-resilient states.
  Arms: Emotional Brain Training (EBT) and Standard of Care (SOC)
Other: Standard addiction counseling and medical therapy — Participants will receive standard counseling (including but not limited to cognitive behavioral therapy, motivational interviewing, etc.), which does not include EBT, in addition to medications for addiction treatment (including but not limited to buprenorphine, naltrexone, bupropion, etc.).

SUMMARY:
The goal of this clinical trial is to determine whether Emotional Brain Training (EBT), a behavioral modification method, can help manage stress and health problems related to addiction. EBT teaches skills to deactivate harmful circuits (automatic reactions) and activate healing circuits to quickly shift mood from negative to positive. Participants in the EBT group will receive focused, intensive instruction on using these skills to rewire unwanted brain circuits, with the aim of achieving lasting improvements in emotional health and quality of life. The study will assess whether EBT is an effective tool when added to standard of care (SOC), which includes medications for addiction treatment (MAT).

Researchers will compare changes in stress, anxiety, and cravings after 8 weeks of EBT plus SOC versus SOC alone.

Participants:

* will either continue receiving standard treatments (SOC) at the Addiction Recovery Clinic (ARC) at SAC Health in San Bernardino
* or receive both EBT and SOC at ARC
* in the SOC group will continue monthly visits at ARC and weekly counseling
* in the EBT plus SOC group will continue monthly visits and weekly counseling at ARC, along with weekly EBT group sessions by telephone
* will complete online assessments at weeks 0, 4, and 8 Upon completion of the study, all participants will resume SOC

DETAILED DESCRIPTION:
Background Information and Rationale Addiction is a neuropsychological disorder defined by a persistent and intense urge to use a drug or engage in a behavior that produces a natural reward, despite significant harm and negative consequences. Repetitive substance use alters brain function, perpetuating craving and weakening self-control, while not completely negating it. Addiction is now recognized as a complex brain disorder influenced by both neurobiological and psychosocial factors. Effective treatment typically combines pharmacological approaches with behavioral interventions, such as cognitive behavioral therapy (CBT), psychotherapy, behavior modification strategies, twelve-step programs, and structured residential care.

Emotional Brain Training (EBT) is a method of self-directed neuroplasticity targeting the neural root causes of addiction, rather than substituting one addiction for another. EBT addresses three primary brain-based contributors to addiction:

1. Replacing self-regulatory failure with optimal brain-based self-regulation, even under stress.
2. Rewiring maladaptive survival and core circuits to become stress resilient.
3. Raising the brain's physiological set point from allostatic to homeostatic, supporting adaptive lifestyle changes and reliance on natural rewards.

The core therapeutic technique of EBT is a structured emotional resiliency process that rewires maladaptive circuits through:

1. Activation of stress-related survival circuits.
2. Emotional processing to shift circuits from allostatic to homeostatic states.
3. Conscious identification of maladaptive expectations.
4. Juxtaposition of adaptive expectations to promote circuit reconsolidation.
5. Delivery of a dopamine release to solidify the rewiring. This process, consistent with reconsolidation research, is repeated until maladaptive drives and responses are eliminated.

EBT uniquely targets brain circuits that control physiology. The same set of skills is applied by clinicians, in peer-to-peer support, and through self-care with mobile app support, enhancing access and scalability. Delivery occurs through small group telephonic sessions using a confidential platform that fosters learning, community, and coaching.

Group sessions are facilitated by licensed health professionals or certified coaches trained in personal and clinical EBT use. Emotional resiliency processes can be completed rapidly, ranging from two to three minutes for self-regulation to approximately twenty minutes for clinician-facilitated trauma rewiring. Practice is further reinforced through brief peer-to-peer sessions and mobile app exercises.

EBT effectiveness has been evaluated in 14 small studies, demonstrating improvements in psychological measures (such as depression, perceived stress, and self-efficacy), behavioral outcomes (including reduced addictive behaviors and increased exercise), and physiological markers (such as blood pressure and BMI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Patient can speak and read English
* Patient who receives regular MAT care at SAC Health
* Patients who have regular and reliable cellular and/or reliable internet connection
* Patients who are willing to spend average of 25 minutes per day and attend weekly group meetings
* Patients willing to actively participate in group sessions
* Opioid use disorder, at least in early remission
* Alcohol use disorder, at least in early remission
* Methamphetamine use disorder, at least in early remission
* Cocaine use disorder, at least in early remission
* Anxiolytic use disorder, at least in early remission
* Cannabis use disorder
* Tobacco use disorder

Exclusion Criteria:

* Age <18 years old
* Patient does not speak or read English
* Patients who do not seek regular MAT care at SAC Health
* Patients with inconsistent or no access to cellular or internet connection
* Any disorder that is uncontrolled
* Any substance use disorder not in at least early remission
* Any patient with complications related to use disorder
* Patients enrolled in the Coachella Valley Rescue Mission patients a part of SAC Health
* Anyone who, in the opinion of the investigators, would be unable to participate in an 8-week trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Level of Stress at 8 weeks | Change between baseline(time of study enrollment) and Study completion (8 weeks).
  Level of stress will be measured by comparing scores from baseline to study completion. Responses will be collected using a 10-item survey assessing perceived stress, administered at enrollment and at eight weeks post-enrollment. Each item uses a 5-point Likert scale ranging from "Never" to "Very Often." Scores will be summed to create a composite stress score, with higher scores indicating greater perceived stress. This measurement evaluates how often participants experience emotional and cognitive responses to stressors such as lack of control, feeling overwhelmed, or being unable to cope.
Changes of Level of Anxiety at 8 weeks | Change between baseline(time of study enrollment) and Study completion (8 weeks).
  Level of anxiety will be assessed using a standardized PROMIS anxiety scale. Participants will complete the survey at baseline and again at the end of the eight-week study period. The survey consists of 8 items rated on a 5-point Likert scale from "Never" to "Always." Items measure frequency of symptoms such as nervousness, tension, and difficulty concentrating due to anxiety. A composite score will be calculated, with higher values reflecting more severe anxiety symptoms.
Change in Levels of Cravings | Change between baseline(time of study enrollment) and Study completion (8 weeks).
  Level of cravings will be measured using selected items from the TAPS (Tobacco, Alcohol, Prescription medication, and other Substance use) assessment tool. Participants will report frequency of use and urges related to substance use at baseline and again at the end of the eight-week period. Responses will be categorized to identify changes in craving intensity and frequency. Increased scores suggest more frequent or intense cravings, while lower scores indicate a reduction in craving-related behaviors or urges.

SECONDARY OUTCOMES:
Change in level of stress (week 4 to 8) | Change between mid-point(week 4) and Study completion (8 weeks).
  Level of stress will be measured at three timepoints: baseline (week 0), midpoint (week 4), and study completion (week 8). Responses will be collected using a 10-item perceived stress scale. Each item is rated on a 5-point Likert scale ranging from "Never" to "Very Often." A composite stress score will be calculated at each timepoint, with higher scores reflecting greater perceived stress. The measure evaluates emotional and cognitive responses to stressors, such as unpredictability, lack of control, and feeling overwhelmed. Changes in stress levels will be tracked across the study duration.
Change in level of anxiety (week 4 to 8) | Change between mid-point(week 4) and Study completion (8 weeks).
  Anxiety will be assessed at baseline, 4 weeks, and 8 weeks using the PROMIS anxiety scale. This 8-item instrument uses a 5-point Likert scale from "Never" to "Always" to evaluate symptoms such as nervousness, tension, and difficulty focusing. A composite anxiety score will be calculated for each assessment point. Higher scores indicate more severe anxiety. Changes will be examined over time to evaluate the trajectory of anxiety symptoms during the intervention.
Change in level of cravings (week 4 to 8) | Change between mid-point(week 4) and Study completion (8 weeks).
  Craving levels will be measured at weeks 0, 4, and 8 using selected items from the TAPS (Tobacco, Alcohol, Prescription medication, and other Substance use) tool. Participants will report frequency of substance use and associated urges. Responses will be used to generate categorical indicators of craving intensity and frequency. Changes across timepoints will be used to determine patterns in craving reduction or escalation throughout the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Addiction Recovery Clinic at SAC Health, San Bernardino, California, United States

IPD SHARING:
Plan to Share IPD: No
Pilot project. Need specifically qualified EBT trainer for this study.

REFERENCES:
- [Background] Mellin L, Fish-dePena LE, Frassetto LA, Mitrovic I. Rewiring the stress response: A new paradigm for health care. Medical Hypothesis 9(1), 2011.
- [Background] Clay SW, Allen J, Parran T. A review of addiction. Postgrad Med. 2008 Jul 31;120(2):E01-7. doi: 10.3810/pgm.2008.07.1802. PMID 18654058
- [Background] Henden E (2017). Addiction, compulsion, and weakness of the will: A dual-process perspective.. In Heather N, Gabriel S (eds.). Addiction and Choice: Rethinking the Relationship. Oxford, UK: Oxford University Press. pp. 116-132
- [Background] "Drugs, Brains, and Behavior: The Science of addiction - Drug misuse and addiction. www.drugabuse.gov. North Bethesda, Maryland: National Institute on Drug Abuse. 13 July 2020. Retrieved 23 December 2021.
- [Background] Nestler EJ. Cellular basis of memory for addiction. Dialogues Clin Neurosci. 2013 Dec;15(4):431-43. doi: 10.31887/DCNS.2013.15.4/enestler. PMID 24459410
- [Background] Heilig M, MacKillop J, Martinez D, Rehm J, Leggio L, Vanderschuren LJMJ. Addiction as a brain disease revised: why it still matters, and the need for consilience. Neuropsychopharmacology. 2021 Sep;46(10):1715-1723. doi: 10.1038/s41386-020-00950-y. Epub 2021 Feb 22. PMID 33619327
- [Result] Ford J, Frassetto L, Mellin L. Emotional Brain Training (EBT) in Subjects after Bariatric Surgery. American Society of Bariatric Surgery, Virginia Beach 8.19.23 abstract - first place.
- See also: website describing EBT — https://www.ebtconnect.net/